CLINICAL TRIAL: NCT01469598
Title: Phase II Study of Docetaxel and Gemcitabine in Previously Treated Metastatic Esophageal Squamous Cell Cancer
Brief Title: Study of Docetaxel and Gemcitabine in Metastatic Esophageal Squamous Cell Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jeeyun Lee, Professor of Medicine, Sungkyunkwan University School of Medicine, Department of Hematology and Oncology, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-03-053
Record Dates: First submitted 2011-11-07; First posted 2011-11-10 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2015-12

CONDITIONS: Metastatic Carcinoma; Recurrent Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Carcinoma; Esophageal Squamous Cell Carcinoma | interventions — Gemcitabine; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gemcitabine/Docetaxel (Experimental): Gemcitabine 1000 mg/m2 IV over 10 mg/m2/min Docetaxel 35 mg/m2 IV over 1hr every 21 days
  Interventions: Drug: Gemcitabine/Docetaxel

INTERVENTIONS:
Drug: Gemcitabine/Docetaxel — Gemcitabine 1000 mg/m2 IV over 10 mg/m2/min Docetaxel 35 mg/m2 IV over 1hr every 21 days

SUMMARY:
Gemcitabine is a novel analog of the nucleoside deoxycytidine that acts via inhibition of DNA synthesis.Docetaxel is a semisynthetic taxane and promotes microtubule assembly and inhibits microtubule depolymerization.

In this study, patients received gemcitabine 900 mg/m2 on days 1 and 8 plus docetaxel 100 mg/m2 on day 8 with G-CSF support every 3 week.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic, or recurrent esophageal squamous cell carcinoma
* Age > 18 years
* ECOG performance status 0 - 2
* At least one measurable lesion(s) by RECIST 1.1 criteria
* Life expectancy ≥ 3 months
* At least one cytotoxic chemotherapy regimen (adjuvant chemotherapy will be considered as one regimen if administered within 6 months from the date of study entry) (upto three prior regimens will be allowed)
* Prior radiotherapy must be completed 2 weeks before study entry.
* Adequate bone marrow function (≥ ANC 1,500/ul, ≥ platelet 100,000/ul, ≥ Hemoglobin 9.0 g/dl)
* Adequate renal function (≤ serum creatinine 1.5 mg/dl or CCr ≥ 50 ml/min)
* Adequate liver function (≤ serum bilirubin 1.5 mg/dl, ≤ AST/ALT x 3 upper normal limit)
* Written informed consent

Exclusion Criteria:

* Evidence of serious gastrointestinal bleeding
* Serious pulmonary conditions/illness (e.g. chronic lung disease with hypoxemia)
* Serious metabolic disease such as severe non-compensated diabetes mellitus
* History of significant neurologic or psychiatric disorders
* Serious uncontrolled intercurrent infections, or other serious uncontrolled concomitant disease
* Pregnant or lactating woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-08; Primary Completion 2014-02 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Response rate | 1years

SECONDARY OUTCOMES:
progression free survival | 1years
overall survival | 1years
Number of Adverse Events | 1years

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung medical Center, Seoul, South Korea